CLINICAL TRIAL: NCT04125550
Title: The Anti-inflammatory and Anti-oxidant Effects of Propofol and Sevoflurane in Children With Cyanotic Congenital Heart Disease
Brief Title: Propofol vs Sevoflurane in Cyanotic Congenital Heart Disease
Acronym: PSI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Feride Karacaer, Associate Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Cyanotic children
Record Dates: First submitted 2019-07-09; First posted 2019-10-14 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Cyanotic Congenital Heart Disease; Pediatric HD
MeSH Terms: interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group P (Experimental): In Group P, 2-3 mg/kg propofol, 5 µg/kg iv fentanyl will be administered for anesthesia induction and 0.6 mg/kg rocuronium will be used as muscle relaxants. 10 mg/kg/h propofol infusion and 5 µg/kg/h fentanyl infusion will be administered.
  Interventions: Drug: Propofol
- Group S (Active Comparator): In Group S, sevoflurane inhalation (2-8%), 5 microgr/kg intravenous (iv) fentanyl will be administered for anesthesia induction and 0.6 mg/kg rocuronium will be used as muscle relaxants. 2% sevoflurane inhalation and 5 µg/kg/h fentanyl infusion will be administered for the maintenance of anesthesia.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — 2-3 mg/kg propofol will be administered for anesthesia induction. 10 mg/ kg/h propofol infusion will be administered for the maintenance of anesthesia.
  Arms: Group P
Drug: Sevoflurane — sevoflurane inhalation (2-8%) will be administered for anesthesia induction. 2% sevoflurane inhalation will be administered for the maintenance of anesthesia.
  Other Names: Sevorane
  Arms: Group S

SUMMARY:
The stress response to surgery compromises a series of humoral, metabolic, or cellular reactions. Cardiac surgery with use of cardiopulmonary bypass (CPB) is a major activator of the systemic inflammatory response (SIRS). Inflammation, resulting in neutrophil activation, plays a central role in the production of reactive oxygen species (ROS). Inflammatory and oxidative reactions may play a role in the more frequent observation of postoperative ventricular dysfunction in patients with cyanotic congenital heart disease (CHD) undergoing surgery. The aim of this study is to compare the anti-inflammatory and anti-oxidant effects of propofol and sevoflurane in children with cyanotic CHD undergoing open heart surgery with CPB.

DETAILED DESCRIPTION:
The stress response to surgery compromises a series of humoral, metabolic, or cellular reactions. Cardiac surgery with use of cardiopulmonary bypass (CPB) is a major activator of the systemic inflammatory response (SIRS). Inflammation, resulting in neutrophil activation, plays a central role in the production of reactive oxygen species (ROS). Neutrophil activation and IRI during CPB plays a central role the production of free radicals. An imbalance between the free radicals and the antioxidant capacity of the body results oxidative stress, which leads to lipid, protein and DNA damage Despite significant refinements over the years, inflammation remain major concerns when using CPB.

SIRS was more prevalent in patients operated for tetralogy of Fallot and cyanotic syndromes. It has been shown that pro-inflammatory cytokines are present in the myocardium of patients with congenital heart disease and concentrations are higher in cyanotic patients than in acyanotic patients. During CPB, more free oxygen radical production occurs in response to reoxygenation after chronic cyanosis. Inflammatory and oxidative reactions may play a role in the more frequent observation of postoperative ventricular dysfunction in patients with cyanotic congenital heart disease (CHD) undergoing surgery.

Propofol has been suggested as a useful adjunct to CPB because of its potential protective effect on the heart mediated by a decrease in ischemia-reperfusion injury and inflammation at clinically relevant concentrations. The anti-inflammatory potential of sevoflurane has been confirmed in several clinical studies, including patients undergoing cardiac surgery with the use of CPB.

The goal of anesthetic management of children with CHD is to ensure an ongoing intraoperative and postoperative cardiovascular stability with attenuation of the stress response and nociceptive stimulation. Postoperative morbidity and mortality may be reduced by anesthetic agents which prevent inflammatory and oxidative reactions. The aim of this study is to compare the anti-inflammatory effects of propofol and sevoflurane in children with cyanotic CHD undergoing open heart surgery with CPB.

34 patients aged 1-10 years undergoing open heart surgery for cyanotic congenital heart disease will be included in the study.Patients will be randomly divided into two groups.

In Group S, sevoflurane inhalation (2-8%), 5 microgr/kg intravenous (iv) fentanyl will be administered for anesthesia induction and 0.6 mg/kg rocuronium will be used as muscle relaxant. 2% sevoflurane inhalation and 5 µg/kg/h fentanyl infusion will be administered for the maintenance of anesthesia.

In Group P, 2-3 mg/kg propofol, 5 µg/kg iv fentanyl will be administered for anesthesia induction and 0.6 mg/kg rocuronium will be used as muscle relaxant. 10 mg/ kg/h propofol infusion and 5 µg/kg/h fentanyl infusion will be administered for the maintenance of anesthesia..

Blood samples were collected at four time points: before operation (T0), after release of the aortic cross-clamp (T1), at the end of the operation (T2), 24 h after the operation (T3). The blood samples were centrifuged at 1,000xg for 15 min and the serum samples were stored at -80 0C until analysis.

Serum interleukin-6 (IL-6) tumor necrosis alpha (TNF-alpha), total anti-oxidant status (TAS) and total oxidant status (TOS) levels will be measured.

In the postoperative period, age-specific SIRS criteria determined by the International Pediatric Sepsis Consensus Conference will be used. Patients will be evaluated for SIRS diagnosis at 6, 12 and 24 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* 1-10 years old
* Patients with cyanotic congenital heart disease undergoing open heart surgery with CPB

Exclusion Criteria:

* Patients with liver or renal dysfunction
* Patients with inflammatory disease
* Patients with hemostatic disorders
* Preoperative use of anti-inflammatory and/or antioxidant drugs

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Interleukin-6 level at postoperative 24.hours | Interleukin-6 level at postoperative 24.hours
  Serum interleukin-6 (IL-6) level will be measured.

SECONDARY OUTCOMES:
Tumor necrosis factor alpha (TNF-alpha) level | Serum TNF-alpha level at postoperative 24.hours
  Serum TNF-alpha level will be measured.
Total anti-oxidant status (TAS) level | Serum TAS level at postoperative 24. hours
  Serum TAS level will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Feri̇de Karacaer, Study Director — Cukurova University
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)